CLINICAL TRIAL: NCT04377633
Title: Impact of an Anesthesia-handover Checklist on Perioperative Outcomes of Elderly Patients Undergoing Major Noncardiac Surgery: A Prospective Before-and-after Study
Brief Title: Anesthesia-handover Checklist and Perioperative Outcomes in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2020-042
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Elderly Patients; Major Surgery; Anesthesia; Adverse Effect; Prevention; Postoperative Complications
Keywords: Elderly patients; Major surgery; Anesthesia handover; Handover checklist; Postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (Sham Comparator): Anesthesia handover during surgery will be performed as usual, i.e., a verbal exchange of pertinent clinical information.
  Interventions: Procedure: Oral handover
- Post-intervention (Experimental): Anesthesia handover during surgery will be performed according to a structured checklist.
  Interventions: Procedure: Checklist handover

INTERVENTIONS:
Procedure: Oral handover — Anesthesia handover during surgery will be performed as usual, i.e., oral exchange of pertinent clinical information.
  Arms: Pre-intervention
Procedure: Checklist handover — Anesthesia handover during surgery will be performed according to a structured handover checklist.
  Arms: Post-intervention

SUMMARY:
With the increasing number of surgical cases, intraoperative handover of anesthesia care is common and inevitable. Verbal handover from one anesthesiologist to another during surgery are being used in many hospitals. However, verbal handover is often an informal, unstructured process during which omissions and errors can occur. It is possible that an improved anesthesia handover may reduce the related adverse events. This study aims to test the hypothesis that use of a well-designed, structured handover-checklist to improve handover quality may decrease the occurrence of postoperative complications in elderly patients undergoing major noncardiac surgery.

DETAILED DESCRIPTION:
It was estimated that more than 9 million patients undergo surgery with a complete anesthesia handover each year worldwide. Verbal handover from one anesthesiologist to another during surgery are being used in many hospitals; and there is no unified patient handover guideline at present.

It is well recognized that the transfer-of-care is a point of vulnerability where valuable patient information can be distorted and omitted. A previous study of the investigators showed that handover of anesthesia care was associated with a higher risk of delirium in elderly patients after major noncardiac surgery. The World Health Organization has included communication during patient care handovers among its top 5 patient safety initiatives.

It is possible that an improved anesthesia-handover protocol may reduce the related adverse events. Many efforts have performed to optimize handover processes. However, handover quality between anesthesiologists has rarely been investigated. The investigators hypothesize that a well-designed, structured handover-checklist will improve handover quality and reduce the occurrence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients (aged 65 years and over);
2. Scheduled to undergo major non-cardiac surgery with an expected duration of at least 2 hours;
3. Requirement of complete handover between anesthesiologists during surgery (initial anesthesiologist no longer returns).

Exclusion Criteria:

1. Preoperative history of schizophrenia, epilepsy, Parkinsonism or myasthenia gravis;
2. Inability to communicate before surgery (coma, profound dementia or language barrier);
3. Craniocerebral injury or neurosurgery;
4. Severe liver dysfunction (Child-Pugh grade C), severe renal dysfunction (requiring dialysis), or expected survival of <24 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1421 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
A composite incidence of all complications within 30 days after surgery. | Up to 30 days after surgery.
  Include organ injury (delirium, acute kidney injury, and myocardial injury) within 3 days and other major complications (class II or higher on Clavien-Dindo classification) within 30 days after surgery.

SECONDARY OUTCOMES:
Intensive care unit admission after surgery. | Up to 30 days after surgery.
  Intensive care unit admission after surgery.
Length of stay in the intensive care unit after surgery. | Up to 30 days after surgery.
  Length of stay in the intensive care unit after surgery.
Incidence of organ injury (delirium, acute kidney injury, and acute myocardial injury) within 3 days after surgery. | Up to 3 days after surgery.
  Delirium is diagnosed with the Confusion Assessment Method. Acute kidney injury is diagnosed according to the KDIGO (Kidney Disease: Improving Global Outcomes) Criteria. Acute myocardial injury is diagnosed according to the serum cardiac tropinin I level.
Incidence of major complications within 30 days after surgery. | Up to 30 days after surgery.
  Major complications are defined as newly occurred conditions that are harmful to patients' recovery and required medical therapy, i.e., class II or higher on the Clavien-Dindo classification.
Length of hospital stay after surgery. | Up to 30 days after surgery.
  Length of hospital stay after surgery.
All-cause mortality within 30 days after surgery. | Up to 30 days after surgery.
  All-cause mortality within 30 days after surgery.

OTHER OUTCOMES:
Pain intensity within 3 days after surgery. | Up to 3 days after surgery.
  Pain intensity is assessed with the Numeric Rating Scale, an 11-point scale where 0=no pain and 10=the worst pain.
Subjective sleep quality within 3 days after surgery. | Up to 3 days after surgery.
  Subjective sleep quality is assessed with the Numeric Rating Scale, an 11-point scale where 0=the best sleep and 10=the worst sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choromanski D, Frederick J, McKelvey GM, Wang H. Intraoperative patient information handover between anesthesia providers. J Biomed Res. 2014 Sep;28(5):383-7. doi: 10.7555/JBR.28.20140001. Epub 2014 Jun 10. PMID 25332710
- [Background] Siddiqui N, Arzola C, Iqbal M, Sritharan K, Guerina L, Chung F, Friedman Z. Deficits in information transfer between anaesthesiologist and postanaesthesia care unit staff: an analysis of patient handover. Eur J Anaesthesiol. 2012 Sep;29(9):438-45. doi: 10.1097/EJA.0b013e3283543e43. PMID 22569028
- [Background] Singh H, Thomas EJ, Petersen LA, Studdert DM. Medical errors involving trainees: a study of closed malpractice claims from 5 insurers. Arch Intern Med. 2007 Oct 22;167(19):2030-6. doi: 10.1001/archinte.167.19.2030. PMID 17954795
- [Background] Arora V, Johnson J, Lovinger D, Humphrey HJ, Meltzer DO. Communication failures in patient sign-out and suggestions for improvement: a critical incident analysis. Qual Saf Health Care. 2005 Dec;14(6):401-7. doi: 10.1136/qshc.2005.015107. PMID 16326783
- [Background] Horwitz LI, Moin T, Krumholz HM, Wang L, Bradley EH. Consequences of inadequate sign-out for patient care. Arch Intern Med. 2008 Sep 8;168(16):1755-60. doi: 10.1001/archinte.168.16.1755. PMID 18779462
- [Background] Hudson CC, McDonald B, Hudson JK, Tran D, Boodhwani M. Impact of anesthetic handover on mortality and morbidity in cardiac surgery: a cohort study. J Cardiothorac Vasc Anesth. 2015 Feb;29(1):11-6. doi: 10.1053/j.jvca.2014.05.018. Epub 2014 Nov 24. PMID 25440620
- [Background] Jones PM, Cherry RA, Allen BN, Jenkyn KMB, Shariff SZ, Flier S, Vogt KN, Wijeysundera DN. Association Between Handover of Anesthesia Care and Adverse Postoperative Outcomes Among Patients Undergoing Major Surgery. JAMA. 2018 Jan 9;319(2):143-153. doi: 10.1001/jama.2017.20040. PMID 29318277
- [Background] Liu GY, Su X, Meng ZT, Cui F, Li HL, Zhu SN, Wang DX. Handover of anesthesia care is associated with an increased risk of delirium in elderly after major noncardiac surgery: results of a secondary analysis. J Anesth. 2019 Apr;33(2):295-303. doi: 10.1007/s00540-019-02627-3. Epub 2019 Feb 28. PMID 30820749
- [Background] Hyder JA, Bohman JK, Kor DJ, Subramanian A, Bittner EA, Narr BJ, Cima RR, Montori VM. Anesthesia Care Transitions and Risk of Postoperative Complications. Anesth Analg. 2016 Jan;122(1):134-44. doi: 10.1213/ANE.0000000000000692. PMID 25794111
- [Background] Kraman SS, Hamm G. Risk management: extreme honesty may be the best policy. Ann Intern Med. 1999 Dec 21;131(12):963-7. doi: 10.7326/0003-4819-131-12-199912210-00010. PMID 10610649
- [Background] Berkenstadt H, Haviv Y, Tuval A, Shemesh Y, Megrill A, Perry A, Rubin O, Ziv A. Improving handoff communications in critical care: utilizing simulation-based training toward process improvement in managing patient risk. Chest. 2008 Jul;134(1):158-62. doi: 10.1378/chest.08-0914. PMID 18628218
- [Background] Wayne JD, Tyagi R, Reinhardt G, Rooney D, Makoul G, Chopra S, Darosa DA. Simple standardized patient handoff system that increases accuracy and completeness. J Surg Educ. 2008 Nov-Dec;65(6):476-85. doi: 10.1016/j.jsurg.2008.06.011. PMID 19059181
- [Background] The Joint Commission releases Improving America's Hospitals: The Joint Commission's Annual Report on Quality and Safety, 2008. Jt Comm Perspect. 2009 Jan;29(1):3, 5. No abstract available. PMID 19368073
- [Background] Ferran NA, Metcalfe AJ, O'Doherty D. Standardised proformas improve patient handover: Audit of trauma handover practice. Patient Saf Surg. 2008 Sep 25;2:24. doi: 10.1186/1754-9493-2-24. PMID 18817559
- [Background] Riesenberg LA, Leitzsch J, Little BW. Systematic review of handoff mnemonics literature. Am J Med Qual. 2009 May-Jun;24(3):196-204. doi: 10.1177/1062860609332512. Epub 2009 Mar 5. PMID 19269930
- [Background] Haynes AB, Weiser TG, Berry WR, Lipsitz SR, Breizat AH, Dellinger EP, Herbosa T, Joseph S, Kibatala PL, Lapitan MC, Merry AF, Moorthy K, Reznick RK, Taylor B, Gawande AA; Safe Surgery Saves Lives Study Group. A surgical safety checklist to reduce morbidity and mortality in a global population. N Engl J Med. 2009 Jan 29;360(5):491-9. doi: 10.1056/NEJMsa0810119. Epub 2009 Jan 14. PMID 19144931
- [Background] Shah AC, Oh DC, Xue AH, Lang JD, Nair BG. An electronic handoff tool to facilitate transfer of care from anesthesia to nursing in intensive care units. Health Informatics J. 2019 Mar;25(1):3-16. doi: 10.1177/1460458216681180. Epub 2016 Dec 1. PMID 29231091
- [Background] Hall M, Robertson J, Merkel M, Aziz M, Hutchens M. A Structured Transfer of Care Process Reduces Perioperative Complications in Cardiac Surgery Patients. Anesth Analg. 2017 Aug;125(2):477-482. doi: 10.1213/ANE.0000000000002020. PMID 28504990
- [Background] Kalkman CJ. Handover in the perioperative care process. Curr Opin Anaesthesiol. 2010 Dec;23(6):749-53. doi: 10.1097/ACO.0b013e3283405ac8. PMID 21037475
- [Background] Catchpole KR, de Leval MR, McEwan A, Pigott N, Elliott MJ, McQuillan A, MacDonald C, Goldman AJ. Patient handover from surgery to intensive care: using Formula 1 pit-stop and aviation models to improve safety and quality. Paediatr Anaesth. 2007 May;17(5):470-8. doi: 10.1111/j.1460-9592.2006.02239.x. PMID 17474955
- [Background] Philibert I, Barach P. The European HANDOVER Project: a multi-nation program to improve transitions at the primary care--inpatient interface. BMJ Qual Saf. 2012 Dec;21 Suppl 1:i1-6. doi: 10.1136/bmjqs-2012-001598. No abstract available. PMID 23173180
- [Background] Wohlauer MV, Arora VM, Horwitz LI, Bass EJ, Mahar SE, Philibert I; Handoff Education and Assessment for Residents (HEAR) Computer Supported Cooperative Workgroup. The patient handoff: a comprehensive curricular blueprint for resident education to improve continuity of care. Acad Med. 2012 Apr;87(4):411-8. doi: 10.1097/ACM.0b013e318248e766. PMID 22361791
- [Background] Arriaga AF, Elbardissi AW, Regenbogen SE, Greenberg CC, Berry WR, Lipsitz S, Moorman D, Kasser J, Warshaw AL, Zinner MJ, Gawande AA. A policy-based intervention for the reduction of communication breakdowns in inpatient surgical care: results from a Harvard surgical safety collaborative. Ann Surg. 2011 May;253(5):849-54. doi: 10.1097/SLA.0b013e3181f4dfc8. PMID 21173696
- [Background] Petrovic MA, Martinez EA, Aboumatar H. Implementing a perioperative handoff tool to improve postprocedural patient transfers. Jt Comm J Qual Patient Saf. 2012 Mar;38(3):135-42. doi: 10.1016/s1553-7250(12)38018-5. PMID 22435231
- [Background] Pugel AE, Simianu VV, Flum DR, Patchen Dellinger E. Use of the surgical safety checklist to improve communication and reduce complications. J Infect Public Health. 2015 May-Jun;8(3):219-25. doi: 10.1016/j.jiph.2015.01.001. Epub 2015 Feb 26. PMID 25731674
- [Background] Gaba DM. Anaesthesiology as a model for patient safety in health care. BMJ. 2000 Mar 18;320(7237):785-8. doi: 10.1136/bmj.320.7237.785. No abstract available. PMID 10720368
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542